CLINICAL TRIAL: NCT01784081
Title: iPC3 - Integrating Palliative Care and Modern Palliative Care Tools Into the Care of Patients With Pancreas Cancer
Brief Title: Integrating Palliative Care and Modern Palliative Care Tools Into the Care of Patients With Pancreas Cancer
Acronym: iPC3
Status: Withdrawn | Type: Observational
Why Stopped: study was closed by PI due to no accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J1270; 90049470 (Other Grant/Funding Number: Ho-Chiang Foundation); NA_00074891 (Other: JHMIRB)
Record Dates: First submitted 2013-01-23; First posted 2013-02-05 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Pancreas Cancer
Keywords: palliative care; decision aid
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Palliative Care; Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- palliative care with iPC3: Palliative care with decision aids will be administered at each palliative care visit.
  Interventions: Other: Palliative care with decision aids

INTERVENTIONS:
Other: Palliative care with decision aids — Participant is followed by the palliative care team, and at each visit, patient will assess their distress and symptoms. Patients facing a treatment decision will receive a Patient Information Program link to review the diagnosis, prognosis, specific benefits and risks with the proposed chemotherapy.

SUMMARY:
The main purpose of this study is to evaluate the acceptance by patients with metastatic pancreas cancer of integrating palliative care with usual cancer treatment. Palliative care intervention will involve use of pancreas cancer-specific decision aides (iPC3)about prognosis, treatment choices, and advance care planning for patients facing a treatment decision as well as symptom assessments. We hypothesize that palliative care consultations with iPC3 will be accepted, symptoms can be diminished, information can be received in a way that improves choices, and that the quality of care can be improved.

DETAILED DESCRIPTION:
* Each patient undergoing treatment at Johns Hopkins for metastatic pancreas cancer will receive palliative care support during their course to include: palliative care consultation early in their treatment course; patient decision aids that give survival, treatment benefits and risks; suggestions to complete such tasks as advance directives, durable power of medical attorney, wills, family and spiritual reviews as recommend by the American Society of Clinical Oncology; and when indicated, transition to hospice.
* Patient will have an iPad for their visit, and a corresponding website to print information.
* Each patient will assess their distress with the Distress thermometer; symptoms with the Condensed Memorial Symptom Assessment Scale and a depression screen. This information will be given to the health care practitioner before the patient visit.
* Patients facing a treatment decision will receive a Patient Information Program link (or paper for those unable to work on the iPad) to review the diagnosis, prognosis, specific benefits and risks with the proposed chemotherapy. This will then give transition "prompts" to encourage thinking about advance directives, durable power of medical attorney, use of hospice, and doing a life review.
* We will also offer a hospice information visit when patient has - in the projection of the team or treating physician - 3 to 6 months to live.
* The palliative care team will meet at least monthly with each of the enrolled patients.
* Participants will be followed for as long as he or she is alive before receiving hospice care.

ELIGIBILITY:
Inclusion Criteria:

* All patients with metastatic pancreas cancer will be eligible, ages 18 and above.
* There is no limit to the amount of prior therapy for metastatic disease.
* Ability to understand and the willingness to sign a written informed consent document and to answer a questionnaire.
* English speakers.

Exclusion Criteria:

* Patients who have tumors other than metastatic pancreas cancer.
* Patients who actively decline participation or who are judged to be in distress before the interview.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic pancreas cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the patients with metastatic pancreas cancer to meet with the palliative care team and to complete symptom assessments. | participants will be followed monthly until referred to hospice or until death, an expected average of 1 year

SECONDARY OUTCOMES:
Changes in symptoms listed in the Memorial Symptom Assessment Scale (condensed version) | participants will be followed monthly until referred to hospice or until death, an expected average of 1 year
  The condensed Memorial Symptom Assessment Scale evaluates 14 symptoms: lack of energy, lack of appetite, pain, dry mouth, weight loss, feeling drowsy, shortness of breath, constipation, difficulty sleeping, difficulty concentrating, nausea, worrying, feeling sad, and feeling nervous.
Changes in the use of wills, living wills, advanced medical directives, durable power of medical attorney and preferred place of death. | 1 year
Changes in hospice referral, use, acceptance, and length of stay, compared to similar patients in the prior 12 months (from retrospective review) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Smith, MD, Principal Investigator — Johns Hopkins Medical Institutions, Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Smith TJ, Temin S, Alesi ER, Abernethy AP, Balboni TA, Basch EM, Ferrell BR, Loscalzo M, Meier DE, Paice JA, Peppercorn JM, Somerfield M, Stovall E, Von Roenn JH. American Society of Clinical Oncology provisional clinical opinion: the integration of palliative care into standard oncology care. J Clin Oncol. 2012 Mar 10;30(8):880-7. doi: 10.1200/JCO.2011.38.5161. Epub 2012 Feb 6. PMID 22312101